CLINICAL TRIAL: NCT07204262
Title: Integrating Longitudinal Biomarker Dynamics With Clinical Features for Prognostic Prediction in Hepatocellular Carcinoma
Brief Title: Trajectory-Based Prognostic Modeling in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Xu Yong, MD (Other)
Responsible Party: Sponsor-Investigator, Xu Yong, MD, Secretary of the Party Committee & Principal Investigator, Shenzhen Third People's Hospital
Organization: Shenzhen Third People's Hospital (Other)
Other Study IDs: KY2024-179
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Molecular Targeted Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed, paraffin-embedded (FFPE) pathological tissue slides from tumor samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced HCC Cohort: This cohort includes patients with advanced hepatocellular carcinoma (HCC) who received systemic therapy with molecular targeted agents (TKIs or anti-VEGF antibodies) and/or PD-(L)1 inhibitors, with or without interventional treatments such as transarterial chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC). Clinical, radiological, and laboratory data were collected retrospectively to evaluate longitudinal biomarker trajectories and construct prognostic models.
  Interventions: Combination Product: Molecular Targeted Therapy (TKI / anti-VEGF antibody) PD-(L)1 Inhibitor Immunotherapy Interventional Therapy (TACE / HAIC)

INTERVENTIONS:
Combination Product: Molecular Targeted Therapy (TKI / anti-VEGF antibody) PD-(L)1 Inhibitor Immunotherapy Interventional Therapy (TACE / HAIC) — Patients in this study received systemic therapy with molecular targeted agents, including tyrosine kinase inhibitors (TKIs) and anti-VEGF antibodies, and/or PD-(L)1 inhibitor immunotherapy. Some patients also received interventional therapies such as transarterial chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC). Treatment regimens, combinations, and sequencing were determined based on physician discretion and patient clinical status. This study focuses on the longitudinal monitoring of biomarkers during these therapies to evaluate their prognostic value and to develop a trajectory-based risk stratification model for advanced hepatocellular carcinoma (HCC).

SUMMARY:
To evaluate whether tracking changes in key blood markers over time, together with clinical features, can improve the prediction of outcomes in patients with hepatocellular carcinoma (HCC). By developing a trajectory-based prognostic model, we aim to provide more accurate risk assessment and support personalized treatment decisions.

DETAILED DESCRIPTION:
This study retrospectively analyzed patients with advanced hepatocellular carcinoma (HCC) who were treated at Shenzhen Third People's Hospital between 2018 and 2024. Eligible participants received systemic therapy with molecular targeted agents or PD-(L)1 inhibitors, with or without interventional procedures such as transarterial chemoembolization (TACE) or hepatic arterial infusion chemotherapy (HAIC).

Clinical, radiological, and laboratory data were collected at baseline and during follow-up. Blood tests were performed at regular intervals, and imaging evaluations with contrast-enhanced CT or MRI were conducted every 6-12 weeks in accordance with standard practice. Demographic information, disease stage, comorbidities, and treatment- or disease-related complications were also recorded.

The study focuses on the analysis of longitudinal biomarker changes, with the aim of developing prognostic models that integrate biomarker trajectories with clinical features. The ultimate goal is to improve dynamic risk stratification and support personalized treatment decisions for patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically or radiologically confirmed HCC;
2. availability of pre- treatment clinical record, radiological and hematological data and more than 2 cycles of post-treatment data;
3. receipt of treatment during the study period;
4. Age rather than 18 years old.

Exclusion Criteria:

1. baseline data missed;
2. Non-primary liver cancer;
3. incomplete follow-up data;
4. Unevaluable lesions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced hepatocellular carcinoma (HCC), age ≥18 years, with complete baseline and follow-up clinical, radiological, and laboratory data who received systemic or interventional therapy. Patients with non-primary liver cancer, missing data, incomplete follow-up, or unevaluable lesions were excluded.
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Objective Progression-Free Survival (PFS) | Up to approximately 3 years
  To analyse the Progression-Free Survival (PFS) of patients

SECONDARY OUTCOMES:
Objective Secondary Clinical Endpoints - Overall Growth Phase (OS) | Up to approximately 3 years
  To analyse the Secondary Clinical Endpoints - Overall Growth Phase (OS) of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yong Xu, Dr, Study Chair — Shenzhen Third People's Hospital
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No